CLINICAL TRIAL: NCT05834166
Title: Effects of Upper Back Strengthening and Postural Correction on Pain, Functional Status and Sleep Quality in Females With Costal Rib Pain in 3rd Trimester of Pregnancy
Brief Title: Effects of Upper Back Strengthening and Postural Correction in Pregnant Females With Costal Rib Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0524
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper back strengthening and Postural correction: (Experimental): Group A performed exercises for 3 weeks. Participants performed upper back strengthening exercises and postural correction exercises for 10 to 15 minutes per session. All exercises were performed for 3 sessions per week for a period of 4 weeks. The re-assessment will be done at the 6th and 9th visits.
  Interventions: Other: Upper back strengthening and Postural correction
- Control group: (No Intervention): Group B: Group B will receive no intervention. Baseline treatment will include soft tissue mobilization, chest muscle stretch, trunk muscle stretch, and diaphragmatic breathing exercises for all patients

INTERVENTIONS:
Other: Upper back strengthening and Postural correction — The treatment protocol will involve upper back strengthening exercises and postural correction exercises 3 times a week for 10 to 15 minutes. Upper back strengthening will involve exercises with light-to-moderate load of free weights (body weight or resistance bands) or with a stability ball. Postural correction will involve maintaining the correct posture.
  Arms: Upper back strengthening and Postural correction:

SUMMARY:
1. Study will be a Non-Randomized clinical trial to check the effects of upper back strengthening and postural correction on pain, functional status and sleep quality in females with costal rib pain in 3rd trimester of pregnancy so that we can devise a treatment protocol for females during pregnancy suffering from costal rib pain. Duration of study was 6 months, Non-probability convenient sampling technique was used, subject following eligibility criteria from Avicenna Hospital were allocated in two groups, baseline assessment was done, Group A participants were given baseline treatment along with upper back strengthening and postural correction exercises, Group B participants were given baseline treatment along with no other specific treatment for 3 weeks. On 6th and 12th day, post intervention assessment was done via, Numeric Pain Rating Scale, Patient Specific Functional Scale and Pittsburgh Sleep Quality Index. 3 sessions per week were given, data was analyzed by using SPSS version 26.

DETAILED DESCRIPTION:
Costal rib pain is very common in pregnancy, especially during the third trimester (weeks 28 to 40). After excluding other serious conditions, this condition can also be diagnosed as intercostal myalgia, costochondritis or muscular strain. There are a lot of causes which can result in costal rib pain such as ribs flaring, hormonal changes, increase in the breast size, inflammation of the ribs cartilage and the stretch on intercostal muscles. It can thus result in pain and discomfort due to which the pregnant females find it difficult to sleep at night and also have functional limitations. The prevalence rate of upper back and costal rib pain in pregnancy is almost 47%. The findings of this study can help physiotherapists to manage the costal rib pain in pregnancy more effectively. This will add valuable knowledge to provide the patients with non-invasive and non-pharmacological options for management of costal rib pain.

There are different structured program with exercises for flexibility, balance and strengthening for the majority of skeletal muscles specifically for the spinal ones, between the 24th and 36th week of pregnancy. Strengthening exercises centered on the trunk reduce pain, improve Quality of life and Physical health in late pregnancy and at two months in the postpartum period. Strengthening exercises also ease the delivery.

Upper back strengthening will involve exercises with light-to-moderate load of free weights (body weight or resistance bands) or with stability ball. Postural correction will involve maintaining the correct posture.

Soft tissue mobilization, chest muscle stretch, trunk muscle stretch and diaphragmatic breathing exercises were incorporated as baseline exercises in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age : 20-40 years Pregnant females in 3rd trimester
* Positive Painful rib syndrome history(6)
* Primigravida

Exclusion Criteria:

* • Tietze syndrome

  * Rib Fractures
  * Rib tip syndrome
  * Slipping Rib Syndrome
  * Any recent trauma (last 6 months)
  * High Risk pregnancy
  * Any bony or soft tissue systemic disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | up to 4 weeks
  The NPRS is a segmented numeric scale in which the respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. NPRS is anchored by terms describing pain severity extremes
Patient Specific Functional Scale | up to 4 weeks
  The PSFS is an activity specific 10 points scale (0-10) in which an initial assessment and a follow up assessment is done. Its average score is 4.5. The rater assigns different activities that are difficult to perform by the patient. It quantifies the activity limitation and measure the functional outcomes after assessment
Pittsburgh Sleep Quality Index | up to 4 weeks
  The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score.. A global PSQI score greater than 5 helps to distinguish good and poor sleepers.

CONTACTS AND LOCATIONS:
Overall Officials: Nayab Naina, MS*, Principal Investigator — Riphah International University
Locations (1):
- Avicenna Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kesikburun S, Guzelkucuk U, Fidan U, Demir Y, Ergun A, Tan AK. Musculoskeletal pain and symptoms in pregnancy: a descriptive study. Ther Adv Musculoskelet Dis. 2018 Nov 19;10(12):229-234. doi: 10.1177/1759720X18812449. eCollection 2018 Dec. PMID 30515249
- [Background] Dunn G, Egger MJ, Shaw JM, Yang J, Bardsley T, Powers E, Nygaard IE. Trajectories of lower back, upper back, and pelvic girdle pain during pregnancy and early postpartum in primiparous women. Womens Health (Lond). 2019 Jan-Dec;15:1745506519842757. doi: 10.1177/1745506519842757. PMID 30991911
- [Background] Watelain E, Pinti A, Doya R, Garnier C, Toumi H, Boudet S. Benefits of physical activities centered on the trunk for pregnant women. Phys Sportsmed. 2017 Sep;45(3):293-302. doi: 10.1080/00913847.2017.1351286. Epub 2017 Jul 27. PMID 28678599
- [Background] Zaruba RA, Wilson E. IMPAIRMENT BASED EXAMINATION AND TREATMENT OF COSTOCHONDRITIS: A CASE SERIES. Int J Sports Phys Ther. 2017 Jun;12(3):458-467. PMID 28593100
- [Background] Germanovich A, Ferrante FM. Multi-Modal Treatment Approach to Painful Rib Syndrome: Case Series and Review of the Literature. Pain Physician. 2016 Mar;19(3):E465-71. PMID 27008303
- [Background] Zaremba S, Mueller N, Heisig AM, Shin CH, Jung S, Leffert LR, Bateman BT, Pugsley LJ, Nagasaka Y, Duarte IM, Ecker JL, Eikermann M. Elevated upper body position improves pregnancy-related OSA without impairing sleep quality or sleep architecture early after delivery. Chest. 2015 Oct;148(4):936-944. doi: 10.1378/chest.14-2973. PMID 25905714
- [Background] Yoo WG. Effect of thoracic stretching, thoracic extension exercise and exercises for cervical and scapular posture on thoracic kyphosis angle and upper thoracic pain. J Phys Ther Sci. 2013 Nov;25(11):1509-10. doi: 10.1589/jpts.25.1509. Epub 2013 Dec 11. PMID 24396221